CLINICAL TRIAL: NCT03831815
Title: Evaluation of Residual Neuromuscular Blockade and of Late Recurarization in the Post Anesthesia Care Unit in Patients Undergoing Videolaparoscopic Cholecystectomy
Status: Completed | Type: Observational
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Renato Santiago Gomez, Doctor, Federal University of Minas Gerais
Other Study IDs: CAAE: 71086417.3.0000.5121
Record Dates: First submitted 2019-02-04; First posted 2019-02-06 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Neuromuscular Block, Residual
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — cisatracurium; Rocuronium

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Grupo C: cisatracurium: Patients were allocated to two groups based on the neuromuscular blocker used by the anesthesiologist who participated in the surgery. In group C, patients received cisatracurium and in group R, rocuronium was administered to patients.
  Interventions: Drug: Cisatracurium
- Grupo R: rocuronium: Patients were allocated to two groups based on the neuromuscular blocker used by the anesthesiologist who participated in the surgery. In group C, patients received cisatracurium and in group R, rocuronium was administered to patients.

INTERVENTIONS:
Drug: Cisatracurium — Patients were allocated to two groups based on the neuromuscular blocker used by the anesthesiologist participating in the surgery. In group C, the patients in whom cisatracurium was given and the R group consisted of the patients in whom rocuronium was administered. It is emphasized that the choice of the neuromuscular blocker was made by the preference and experience of the anesthesiologist of the case and not by randomization or lottery of the patients.
  Other Names: Rocuronium
  Groups: Grupo C: cisatracurium

SUMMARY:
Neuromuscular blockade is essential to provide optimal conditions for tracheal intubation and also to facilitate the performance of surgeries involving mainly the abdominal cavity. The introduction of neuromuscular blockers in clinical practice optimized the execution of mechanical ventilation. Since the use of these drugs, increased intercurrences such as prolonged muscle paralysis and respiratory complications have been observed, resulting in unfavorable outcomes with residual neuromuscular blockade and delayed recurrence due to the occurrence of these complications. The present study aims to evaluate the incidence of residual neuromuscular blockade and late recurarization in the post-anesthetic recovery room in patients submitted to videolaparoscopic cholecystectomy.

DETAILED DESCRIPTION:
This is an observational and prospective study in which patients aged 18-50 years classified as ASA (American Society of Anesthesiologists) I and II, body mass index below 35 and who will undergo cholecystectomy will be included. Patients will be allocated to two groups based on the neuromuscular blocker used by the anesthesiologist who participates in the surgery, ie in group C patients will participate in the administration of cisatracurium and the group R will consist of the patients in whom rocuronium was administered. General anesthesia and assessment of muscle function will be performed by measuring the four-stimulus sequence (SQE) / train of four (TOF) at pre-established times. A residual neuromuscular block is considered to be the patient presenting the value of the four-stimulus sequence of T4 / T1 of less than 0.9.

ELIGIBILITY:
Inclusion Criteria:

* Patients submitted to videolaparoscopic cholecystectomy under balanced general anesthesia. ASA (American Society of Anesthesiologists) patients, class I and II, age group of 18 to 50 years, body mass index below 35.

Exclusion Criteria:

* Patients ASA III or higher; ASA II patients with respiratory comorbidities. Patients with neuromuscular diseases or severe renal or hepatic diseases. Patients submitted to total venous anesthesia. Patients with body temperature below 36 ° C. Replication of the neuromuscular blocker. Use of drugs that accentuate neuromuscular blockade such as calcium channel blockers, inorganic ions (Mg ++, Li ++), aminoglycoside antibiotics, halogenated anesthetics (except sevoflurane), local anesthetics (except lidocaine), benzodiazepines and opioids (except morphine or remifentanil) .

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients of both sexes and who underwent videolaparoscopic cholecystectomy under balanced general anesthesia. ASA (American Society of Anesthesiologists) patients, class I and II, age group of 18 to 50 years, body mass index below 35.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2018-05-18 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
Residual Neuromuscular Blockade | Immediate postoperative period in the post anesthetic recovery room.
  The patient who presented the value of the sequence of four T4 / T1 stimuli of less than 0.9 was considered to have residual neuromuscular block.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Minas Gerais, Faculdade de Medicina, Departamento de Cirurgia., Belo Horizonte, Minas Gerais, Brazil